CLINICAL TRIAL: NCT03562637
Title: The GLORIA Study: A Phase 3, Randomized, Open-Label Study of the Anti-Globo H Vaccine Adagloxad Simolenin (OBI-822)/OBI-821 in the Adjuvant Treatment of Patients With High Risk, Early Stage Globo H-Positive Triple Negative Breast Cancer
Brief Title: Study of Adagloxad Simolenin (OBI-822)/OBI-821 in the Adjuvant Treatment of Patients With Globo H Positive TNBC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: OBI Pharma, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBI-822-011
Record Dates: First submitted 2018-06-06; First posted 2018-06-19 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Triple Negative Breast Cancer
Keywords: Neoadjuvant chemotherapy; Adjuvant chemotherapy; TNBC
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Adagloxad simolenin + OBI-821 in conjunction with SOC (Experimental): Participants will be administered adagloxad simolenin combined with OBI-821 for up to a total of 21 subcutaneous injections over a period of 100 weeks.
  Patient will also receive standard of care (SOC) treatment.
  Interventions: Biological: adagloxad simolenin combined with OBI-821; Device: Globo H IHC Assay; Other: Standard of care treatment
- Standard of Care treatment (Active Comparator): Study visit intervals will be identical to those in Arm 1.
  Patient will receive standard of care (SOC) treatment.
  Interventions: Device: Globo H IHC Assay; Other: Standard of care treatment

INTERVENTIONS:
Biological: adagloxad simolenin combined with OBI-821 — In the neoadjuvant and adjuvant phases of the study for a total of 100 weeks; subcutaneously injections.
  Arms: Adagloxad simolenin + OBI-821 in conjunction with SOC
Device: Globo H IHC Assay — The Globo H IHC assay will be used to identify eligible patients who may clinically benefit from the OBI-822 treatment, defined by Globo H expression.
Other: Standard of care treatment — Standard of care treatment consisting of observation alone, adjuvant capecitabine or platinum monotherapy over a 100 week period.

SUMMARY:
The GLORIA study is a Phase III, randomized, open-label study to prospectively evaluate the efficacy and safety of adagloxad simolenin (OBI 822)/OBI-821 in the adjuvant treatment of patients with high risk, early stage Globo-H Positive TNBC.

ELIGIBILITY:
Inclusion Criteria:

* Documented radiographic and histopathologic confirmed primary localized invasive breast cancer.
* Histologically documented TNBC (estrogen receptor negative [ER-]/progesterone receptor negative [PR-]/human epidermal growth factor 2 negative [HER2-]) defined as ER-negative and PR-negative (≤5% positive cells stain by IHC for both ER and PR), and negative HER2/neu- status, confirmed on tumor sample.
* HER2/neu negative will be defined as one of the following criteria:

  * IHC 0 or 1+
  * Single-probe average HER2 gene copy number of <6 signals/nucleus
  * Dual-probe fluorescent in-situ hybridization (FISH) HER2/neu chromosome 17 (CEP17) non-amplified ratio of <2
* Globo H IHC H-score ≥15 from the residual primary site/or lymph node (if primary site is not available) tumor obtained at time of definitive surgery or initial diagnosis (only if surgical tumor sample is not available). Globo H expression will be determined during pre-screening by Central lab. Instructions for submission of slides/tumor tissue blocks are provided in the protocol and study Lab Manual.
* No evidence of metastatic disease in chest, abdomen and pelvis by CT or other adequate imagining during the Screening Phase. Imaging within 3 months prior to randomization is acceptable as baseline scan. Bone scans and imaging of the brain at screening is optional, and should be symptom directed.
* High risk patients with no evidence of disease after completing standard treatment and meeting ONE of the following criteria:

  * Neoadjuvant chemotherapy followed by definitive surgery: Residual invasive disease following neoadjuvant chemotherapy defined as: A contiguous focus of residual invasive cancer in the surgical breast specimen measuring ≥1 cm in diameter and/or with residual invasive cancer in at least one axillary node (micrometastases or macrometastases), as determined by local pathology review.
  * Definitive surgery followed by adjuvant chemotherapy: Pathological Prognostic Stage IIB, Stage IIIA , Stage IIIB, or Stage IIIC disease according to the 8th edition of the American Joint Committee on Cancer (AJCC) Cancer Staging Manual.
* Must have completed at least 4 cycles of a standard taxane and anthracycline-based multi-agent chemotherapy regimen (or a taxane-only regimen if the patient is ineligible for anthracycline treatment) either in the neoadjuvant or adjuvant setting (e.g., National Comprehensive Cancer Network recommended regimens):.

  * Randomization must occur (a) within 16 weeks after definitive surgery and radiation therapy (if radiation therapy administered) in patients who received neoadjuvant multiagent chemotherapy or, (b) for patients receiving adjuvant multiagent chemotherapy (not including capecitabine, immune checkpoint inhibitor), within 16 weeks after the completion of the adjuvant multiagent chemotherapy and radiation therapy (if radiation therapy administered). Note: patients may be randomized and initiate study treatment concurrent with adjuvant SOC therapy (observation, capecitabine, immune checkpoint inhibitor ± capecitabine).
* Randomization must occur (a) within 16 weeks after definitive surgery and radiation therapy (if radiation therapy administered) in patients who received neoadjuvant multiagent chemotherapy or, (b) for patients receiving adjuvant multiagent chemotherapy (not including capecitabine, immune checkpoint inhibitor), within 16 weeks after the completion of the adjuvant multiagent chemotherapy and radiation therapy (if radiation therapy administered). Note: patients may be randomized and initiate study treatment concurrent with adjuvant SOC therapy (observation, capecitabine, immune checkpoint inhibitor ± capecitabine).
* All treatment-related toxicities resolved to Grade <1 on National cancer institute Common Terminology Criteria for Adverse Events (NCI-CTCAE version 5.0) criteria (except hair loss and ≤Grade 2 neuropathy, which are acceptable).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Females must be either of non-childbearing potential, i.e., surgically sterilized (have documented sterilization, bilateral oophorectomy/salpingectomy at least 3 months before the start of the trial and/or hysterectomy), or one year postmenopausal; or if of childbearing potential must have a negative pregnancy test (urine or serum) at screening.
* Males and females of childbearing potential and their partners must be willing to use effective contraception during the entire Treatment Phase and for at least 4 weeks (28 days) after the last dose of study treatment.
* Adequate hematological, hepatic and renal function as defined below:

  * Absolute neutrophil count (ANC) ≥1,500/µL
  * Platelets ≥75,000/µL
  * Hemoglobin ≥8.5g/dL
  * Serum creatinine ≤1.5 × upper limit of normal (ULN) or calculated creatinine clearance ≥55 mL/min for subjects with creatinine levels >1.5 × institutional ULN (glomerular filtration rate can also be used in place of creatinine or creatinine clearance may be calculated per institutional standard)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 × ULN
  * Alkaline Phosphatase (ALP) ≤2.5 × ULN
  * Serum total bilirubin ≤1.5 × ULN (unless Gilbert's disease is documented)
* Consent to participate with a signed and dated Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved patient informed consent for the study prior to beginning any specific study procedures.
* Ability to understand and willingness to complete all protocol required procedures.

Exclusion Criteria:

* Local recurrence of or previous history of ipsilateral or contralateral invasive breast cancer within 10 years prior to randomization [for synchronous tumors see Exclusion criteria #3]
* Definitive clinical or radiologic evidence of metastatic disease
* Synchronous bilateral breast cancer, unless both tumors are confirmed as TNBC.
* Have received any anti-cancer vaccines
* Concomitant treatment with anticancer therapy other than adjuvant SOC therapy (capecitabine; immune checkpoint inhibitor), or other investigational therapy, if expected during the study
* A history of other malignancies (except appropriately treated melanoma in situ, non melanoma skin carcinoma, carcinoma in situ of the uterine cervix, follicular or papillary thyroid cancer or other non-breast malignancies with a similar outcome to those mentioned above) within 5 years prior to randomization.
* Have any active autoimmune disease or disorder that requires systemic immunosuppressive/immunomodulatory therapy. NOTE: Autoimmune diseases that are confined to the skin (e.g., psoriasis) that can be treated with topical steroids alone are allowed during the study.
* Oral/parenteral corticosteroid treatment (>5 mg/day of prednisone/equivalent), within 2 weeks prior to randomization or anytime during the study. NOTE: inhaled steroids for treatment of asthma; and topical steroids are allowed during the study.
* Any known uncontrolled concurrent illness that would limit compliance with study requirements, including but not limited to ongoing or active infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric disorders, or substance abuse.
* Any known hypersensitivity to active/inactive ingredients in the study drug formulation or known severe allergy or anaphylaxis to fusion proteins.
* Prior receipt of a glycoconjugate vaccine for cancer immunotherapy.
* Known history or positive for human immunodeficiency virus (HIV positive), unless on effective anti-retroviral therapy with undetectable viral load within 6 months of therapy (note: HIV testing not required for study entry).
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection prior to randomization. Patients who have completed curative therapy and have undetectable viral load for HCV are eligible. For patients with evidence of chronic HBV infection, the HBV viral load must be undetectable on suppressive therapy. (note: HBV/HCV testing is not required for study entry).
* Any condition, including significant diseases and/or laboratory abnormalities that would place the patient at unacceptable risk for study participation.
* Currently pregnant or breastfeeding women.
* Currently participating in or has participated in a breast cancer therapeutic clinical trial within 4 weeks (28 days) prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Measuring the effect of adagloxad simolenin (OBI-822)/OBI-821 treatment on improving invasive disease free survival (IDFS) in the study population. | 5 years
  The outcome measure of the study is IDFS, defined by the STEEP system as the first occurrence of the time from the date of randomization to the date of first invasive disease recurrence (local, regional or distant), the date of secondary primary invasive cancer (breast or not), or the date of death from any cause.

SECONDARY OUTCOMES:
Measuring the impact of adagloxad simolenin (OBI-822)/OBI-821 treatment in the study population on Overall Survival (OS). | 7 years
  OS is defined as the time from randomization to date of death from any cause
Measuring the impact of adagloxad simolenin (OBI-822)/OBI-821 treatment in the study population on Quality of Life (QoL). | 7 years
  QoL defined as time to definitive deterioration in Health-related Quality of Life (HRQOL) using the global health status/QoL scale from European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) and the European Quality of Life 5 Dimensions 5 Levels (EQ-5D-5L). QoL baseline established at randomization.
  Definitive deterioration defined as a 5% worsening relative to baseline in the HRQOL scale score from EORTC QLQ-C30 questionnaires with no subsequent improvement above threshold, scored with the EORTC QLQ-C30 v3.0 Scoring Manual. The EQ-5D-5L questionnaire assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, rated by the patient. It is a standardized measure of health status to provide a simple, generic measure of health for clinical and economic appraisal. 28 questions have a 4 point scale: not at all(1) to very much(4). 2 questions have a 7-point scale: very poor (1) to excellent(7).
Measuring the impact of adagloxad simolenin (OBI-822)/OBI-821 treatment in the study population on Breast cancer-free interval (BCFI). | 7 years
  BCFI is defined by the STEEP system as the first occurrence of the time from the date of randomization to the date of the first invasive disease recurrence (local, regional or distant), the date of ductal carcinoma in situ (ipsilateral or contralateral), or the date of death from breast cancer
Measuring the impact of adagloxad simolenin (OBI-822)/OBI-821 treatment in the study population on Distant disease-free survival (DDFS). | 7 years
  DDFS is defined by the STEEP system as the first occurrence of the time from the date of randomization to the date of the first distant disease recurrence, the date of the second primary invasive cancer (non-breast), or the date of death from any cause
Incidence and severity of adverse events (AEs) [Time Frame: AEs will be noted as it occurs, with a timeframe from beginning of randomization to 4 weeks after last dose of study treatment.] | 2 years
  Adverse Events will be graded and recorded by investigators per National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Hope Rugo, MD, Study Chair — University of California, San Francisco
Locations (128):
- United States (12):
  - Moores UCSD Cancer Center, La Jolla, California
  - Kaiser Permanente Medical Center, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Centre, San Francisco, California
  - Miami Cancer Institute, Miami, Florida
  - University of Chicago Medical, Chicago, Illinois
  - University of Maryland Greenbaum Comprehensive Cancer Center, Baltimore, Maryland
  - Henry Ford Medical Center, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Bons Secours St. Francis Medical Oncology Center, Midlothian, Virginia
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Australia (9):
  - Westmead Hospital, Westmead, New South Wales
  - Cancer Care Service, Hervey Bay Hospital, Urraween, Queensland
  - Victoria Breast & Oncology Care, East Melbourne, Victoria
  - Cabrini Malvern, Malvern, Victoria
  - Breast Cancer Research Centre, Nedlands, Western Australia
  - St Vincent's Hospital Sydney, Darlinghurst
  - Gosford Hospital, Gosford
  - St John of God Murdoch Hospital, Murdoch
  - Eastern Health - Maroondah Hospital, Ringwood East
- Brazil (25):
  - Suporte Nutricional e Quimioterapia, Fortaleza, Ceará
  - Centro de Avaliacao de Medicamentos e Especialidades de Pesquisa, Serra, Espírito Santo
  - Hospital Sao Rafael, Salvador, Estado de Bahia
  - Instituto Mario Penna, Belo Horizonte, Minas Gerais
  - Maternidade e Cirurgia Nossa Senhora do Rocio, Campo Largo, Paraná
  - Hospital das Clinicas - Universidade Federal do Parana, Curitiba, Paraná
  - Centro de Tratamento Oncologico LTDA - CTO, Belém, Pará
  - Hospital do Capibaribe, Recife, Pernambuco
  - Real Hospital Portugues de Beneficencia de Pernambuco, Recife, Pernambuco
  - Centro de Pesquisa Vencer & Oncolinca, Teresina, Piauí
  - Hospital de Clinicas de Porto Alegre, Barretos, Rio Grande do Sul
  - Oncosite-Centro de Pesquisa Clinica em Oncologia, Ijuí, Rio Grande do Sul
  - Hospital Escola da Universidade Federal de Pelotas, Pelotas, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Pontificia Universidade Catolica do Rio Grande do Sul (PUCRS) - Hospital Sao Lucas, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor Amazonia, Porto Velho, Rondona
  - Centro Oncologico de Roraima, Boa Vista, Roraima
  - Clinica Supera, Chapecó, Santa Catarina
  - Clinica de Neoplasias Litoral - Itajai, Itajaí, Santa Catarina
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho de Jau, Jaú, São Paulo
  - Centro de Pesquisa Clinica em Hematologia e Oncologia, Santo André, São Paulo
  - Clinicia de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria, São Paulo, São Paulo
  - Instituto Brasileiro de Controle do Cancer, São Paulo, São Paulo
  - Instituto do Cancer do Estado de San Paulo, São Paulo, São Paulo
- China (17):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Cancer Institute and Hospital, Beijing
- Queen Mary Hospital, Hong Kong, Hong Kong
- Mexico (10):
  - Clinica Oncor - Centro de Infusion e Investigacion Oncologia de Satillo, Saltillo, Coahuila
  - Instituto Nacional de Cancerologia, Mexico City, Del Tialpan
  - Investigacion Biomedica para el Desarrollo de Farmacos, Zapopan, Jalisco
  - Sociedad Administradora de Servicios de Salud S.C., Morelia, Michoacán
  - Centro Medico Zambrano Hellion, San Pedro Garza García, Nuevo León
  - Centro Oncologico Estatal Instituto de Seguridad Social del Estado de Mexico y Municipios, Toluca, State of Mexico
  - Investigacion Biomedica para el Desarrollo de Farmacos, S.A. de. C.V, Aguascalientes
  - Centro Estatal de Cancerologia, Chihuahua City
  - Icaro Investigaciones en Medicina S.A. de C.V., Chihuahua City
  - Scientia Investigacion Clinica S.C., Chihuahua City
- Peru (5):
  - Instituto Nacional de Enfermedades Neoplasicas, Lima, Surquillo
  - Instituto Regional de Enfermedades Neoplasicas del Sur, Arequipa
  - Hospital Nacional Edgardo Rebagliati Martins, Unidad de Investigacion de Oncologia Medica, Lima
  - Unidad de Investigacion - Oncologia Medica Clinica San Felipe, Lima
  - Hospital Maria Auxiliadora, Lima
- Poland (6):
  - University Clinical Centre - Hospital, Teaching Dept of Oncology and Radiotherapy, Gdansk
  - Independent Public Healthcare Facility University Hospital in Cracow, Krakow
  - Contemporary Therapy Centre, Lodz
  - Polish Mother's Memorial Hospital Research Instistute, Lodz
  - Central Teaching Hospital of the MOI in Warsaw, Warsaw
  - Maria Sklodowska-Curie National Institute of Oncology, Warsaw
- Russia (13):
  - Nat. Research Mordovia State University, Saransk, Respublika Mordoviya
  - SBIH of Arkhangelsk region "Arkhangelsk Clinical Oncological Dispensary", Arkhangelsk
  - Krasnoyarsk Territorial Clinical Oncology Center named after A.I. Kryzhanovsky, Krasnoyarsk
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow
  - SBIH of Moscow city "Moscow city oncology hospital №62" of Moscow Healthcare department, Moscow
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - Orenburg Regional Clinical Oncological Center, Orenburg
  - N.N. Petrov National Medical Research Center of Oncology, Pesochnyy
  - LLC Medaid, Saint Petersburg
  - SPb SBIH "City Clinical Oncological Dispensary", Saint Petersburg
  - Klinika Luch, Ltd., Saint Petersburg
  - SBHI "Volgograd Regional Oncology Dispensary #3", Volzhskiy
  - SBIH of Yaroslavl region "Regional Clinical Oncological Hospital", Yaroslavl
- South Africa (3):
  - Netcare Milpark Hospital, Johannesburg, Gauteng
  - Wits Clinical Research, a division of Wits Health Consortium (Pty) Ltd, Johannesburg, Gauteng
  - Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
- South Korea (9):
  - Dong-A University Hospital, Busan
  - National Cancer Center, Goyang-si
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
- Taiwan (9):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation Linkou, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Tri-Service General Hospital, Taipei
- Ukraine (9):
  - Dnipropetrovsk Medical Academy of the Ministry of Health of Ukraine, Dnipro
  - City Clinical Hospital #4, Dnipro
  - CI Transcarpathian Cl Onc Center Dep of Surgery#1 SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - CI of Healthcare Regional Clinical Specialized Dispensary of the Radiation Protection, Kharkiv
  - CI of Kherson Reg Council Kherson Regional Oncologic Dispensary, Kherson
  - Medical Center of Vision Partner, Kyiv
  - Medical Center Verum, Kyiv
  - Kyiv Сity Clinical Oncological Center, Kyiv
  - CI Reg. Oncol. Dispanser, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorodetska I, Samusieva A, Lahuta T, Ponomarova O, Socha O, Kozeretska I. Exploring New Frontiers: Alternative Breast Cancer Treatments Through Glycocalyx Research. Breast J. 2025 May 22;2025:9952727. doi: 10.1155/tbj/9952727. eCollection 2025. PMID 40443562
- [Derived] Rugo HS, Cortes J, Barrios CH, Cabrera P, Xu B, Huang CS, Kim SB, Melisko M, Nanda R, Pienkowski T, Rapoport BL, Schwab R. GLORIA: phase III, open-label study of adagloxad simolenin/OBI-821 in patients with high-risk triple-negative breast cancer. Future Oncol. 2022 Oct 21. doi: 10.2217/fon-2022-0812. Online ahead of print. PMID 36268941